CLINICAL TRIAL: NCT02330198
Title: Evidence for Validity and Reliability of the Finnish Version of the Foot and Ankle Ability Measure
Brief Title: Validation of the Foot and Ankle Ability Measure Tool in Finnish
Acronym: FAAM-Fi
Status: Completed | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: T181/2014
Record Dates: First submitted 2014-12-30; First posted 2015-01-01 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-11

CONDITIONS: Ankle Sprain
Keywords: self-reported outcome instrument
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to validate the Foot and Ankle Ability Measure in Finnish.

DETAILED DESCRIPTION:
The aim of this study is to translate and adapt The Foot and Ankle Ability Measure tool (FAAM) in Finnish language and to evaluate the validity and reliability of the Finnish version of the Foot and ankle ability measure tool (FAAM-Fi).

This study is prospective. It is done by interviewing the patients to gather self-reported information of about their ability to perform different activities of daily living and sports. The study has no consequence to the patients, nor to the treatment aimed to solve the problem. This study includes cross-cultural adaptation of the FAAM to Finnish language and validation of the Finnish version of the FAAM.

The forward translation will be done with the method of used by the American Association of Orthopedic Surgeons (AAOS) Outcomes Committee. Two native Finnish-speakers and fluent in English translators, T1 and T2, translate the original version of the FAAM to Finnish language. T1 is aware of the items being examined in in the questionnaire being translated, but not a healthcare professional. T2 is so called naïve translator. A synthesis of T1 and T2 versions, T-12, is conducted under the supervision of a medical linguistic methodologist. The T-12 version is translated back to English by two native, English as their mother tongue speaking translators BT1 and BT2, neither aware nor informed of the items explored nor with medical background.

An expert committee (the medical linguistic professional, the investigator as an orthopedic specialist and the translators) consolidate all the versions and consider the pre-final version of the questionnaire. The expert committee will be in close contact with developers.

The pre-final version is pre-tested with 40 persons with foot and ankle disorders. They will complete the questionnaire and will be interviewed about the meaning of the questions and the response in order to ensure that the adapted version is retaining its equivalence in an applied situation. Possible missing responses are looked for. The last step is submitting the final version, the FAAM-Fi and all the written reports to the committee keeping track of the translated version and the developers of the final version.

Process for validating the FAAM-Fi includes testing it for reliability, validity and its responsiveness. 80 patients receiving either conservative or operative treatment for foot and ankle disorders are recruited from Turku University Hospital and Physiotherapy Consults, Helsinki. 40 patients are treated operatively and 40 conservatively.

40 patients who will receive operative treatment at the Turku University Hospital Foot and ankle unit are asked to answer the questions of the Finnish version of the FAAM, the modified AOFAS foot and ankle scale and the 15-D instrument by a paper or by an electrical version. At the outpatient clinics of Turku University Hospital and Physiotherapy Consults Helsinki 40 foot and ankle patients who will get physiotherapy fill in these forms. 20 of these patients are recruited from Turku University Hospital and 20 from Physiotherapy Consults Helsinki. Those patients who will be treated operatively fill in the questionnaires at the preoperative interview and in the morning of the surgery. The diagnoses are written down as well as the procedures of the operated patients. The patients will re-fill the questionnaires again at the post-operative control at 3 months.

As this is an interview study there will be no randomizing or blinding.

The study will start in October 2014 and the required information should be gathered in six months. Statistical analysis and first results should be ready in June 2015.

Source population is foot and ankle patients at the outpatient clinic of Artro process of the Turku University Hospital and Physiotherapy Consults, Helsinki.

Number of subjects will be 80.

Test-retest repeatability is evaluated statistically by the agreement of repeated tests. Cronbach´s coefficient alpha is calculated to assess internal consistency. Content validity is assessed by floor and ceiling effects. Criterion validity is tested by correlation to the modified AOFAS foot and ankle scale and 15-D. Construct validity is assessed by creating five hypotheses for convergent validity and one for discriminate. Responsiveness is assessed by calculating the effect size and the standardized effect mean.

All data for this study is collected from patient files and hospitals´ electronic patient registry (Artux, BCB Medical Finland). All data is stored and secured in a specific electronic study subject register. Paper data is stored in a locker in the principal investigators office room at the Turku University Hospital. Patient data is accessible to investigators only.

ELIGIBILITY:
Inclusion Criteria:

* Foot and ankle patients who will receive either conservative or operative treatment will be included. Mother language of the patients is Finnish.

Exclusion Criteria:

* Age under 18 or denial of the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 40 patients who will receive operative treatment at the Turku University Hospital Foot and ankle unit, At the outpatient clinics of Turku University Hospital and Physiotherapy Consults Helsinki 40 foot and ankle patients who will get physiotherapy
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2015-03; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Modified American Orthopaedic Foot & Ankle Society (AOFAS) hindfoot score | 3 months

SECONDARY OUTCOMES:
15 D instrument questionnaires | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jaana Koski, PhT, Principal Investigator — physiotherapist; Jukka Kangas, PhT, Principal Investigator — physiotherapist
Locations (1):
- Turku University Hospital Orthopedics department, Turku, Turku, Finland

REFERENCES:
- [Background] Beaton DE, Bombardier C, Guillemin F, Ferraz MB. Guidelines for the process of cross-cultural adaptation of self-report measures. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3186-91. doi: 10.1097/00007632-200012150-00014. No abstract available. PMID 11124735
- [Background] Beaton DE, Schemitsch E. Measures of health-related quality of life and physical function. Clin Orthop Relat Res. 2003 Aug;(413):90-105. doi: 10.1097/01.blo.0000079772.06654.c8. PMID 12897600
- [Background] Guillemin F, Bombardier C, Beaton D. Cross-cultural adaptation of health-related quality of life measures: literature review and proposed guidelines. J Clin Epidemiol. 1993 Dec;46(12):1417-32. doi: 10.1016/0895-4356(93)90142-n. PMID 8263569
- [Result] Borloz S, Crevoisier X, Deriaz O, Ballabeni P, Martin RL, Luthi F. Evidence for validity and reliability of a French version of the FAAM. BMC Musculoskelet Disord. 2011 Feb 8;12:40. doi: 10.1186/1471-2474-12-40. PMID 21303520
- [Result] Carcia CR, Martin RL, Drouin JM. Validity of the Foot and Ankle Ability Measure in athletes with chronic ankle instability. J Athl Train. 2008 Apr-Jun;43(2):179-83. doi: 10.4085/1062-6050-43.2.179. PMID 18345343
- [Result] Mazaheri M, Salavati M, Negahban H, Sohani SM, Taghizadeh F, Feizi A, Karimi A, Parnianpour M. Reliability and validity of the Persian version of Foot and Ankle Ability Measure (FAAM) to measure functional limitations in patients with foot and ankle disorders. Osteoarthritis Cartilage. 2010 Jun;18(6):755-9. doi: 10.1016/j.joca.2010.03.006. Epub 2010 Mar 23. PMID 20338253
- [Result] Martin RL, Irrgang JJ, Burdett RG, Conti SF, Van Swearingen JM. Evidence of validity for the Foot and Ankle Ability Measure (FAAM). Foot Ankle Int. 2005 Nov;26(11):968-83. doi: 10.1177/107110070502601113. PMID 16309613
- [Result] Nauck T, Lohrer H. Translation, cross-cultural adaption and validation of the German version of the Foot and Ankle Ability Measure for patients with chronic ankle instability. Br J Sports Med. 2011 Aug;45(10):785-90. doi: 10.1136/bjsm.2009.067637. Epub 2009 Dec 2. PMID 19955163